CLINICAL TRIAL: NCT06367270
Title: The Application of Pressured Intraperitoneal Aerosol Chemotherapy (PIPAC) for Peritoneal Surface Malignancies
Acronym: PIPAC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. WONG, Yu Hong Ian, Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 23-361
Record Dates: First submitted 2024-04-10; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Peritoneal Metastases
Keywords: Pressured Intraperitoneal Aerosol Chemotherapy (PIPAC); Peritoneal metastases; Oxaliplatin; Intraperitoneal chemotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PIPAC (Experimental)
  Interventions: Drug: Pressured Intraperitoneal Aerosol Chemotherapy

INTERVENTIONS:
Drug: Pressured Intraperitoneal Aerosol Chemotherapy — PIPAC cycles will be scheduled every 6-8 weeks and 2 weeks after the last systemic chemotherapy administration. The bidirectional program for the combination of intraperitoneal and systemic chemotherapy is designed as follows: systemic chemotherapy followed by PIPAC two weeks later, followed by a one-week interval, and then systemic chemotherapy once again until three PIPAC cycles have been completed. Up to a one-week delay in returning to systemic chemotherapy after PIPAC and vice versa were considered acceptable. Systemic drug choice was based on previous chemotherapy exposure and the medical oncologists' decision. The study ends after the 3rd cycle of PIPAC.
  Other Names: PIPAC

SUMMARY:
Pressurized intraperitoneal aerosol chemotherapy (PIPAC) is a novel minimally invasive drug delivery system for patients with peritoneal metastases (PM). It has been considered as a safe and feasible palliative treatment alternative proven by previous phase I studies. Currently available evidence on feasibility, efficacy and tolerability in Asian populations is limited. In this open-label, single-arm, monocentric clinical trial, investigators aim to evaluate the therapeutic efficacy and complications of PIPAC with oxaliplatin as an alternative on patients of unresectable colorectal cancer with PM and doxorubicin and cisplatin on patients of unresectable gastric and pancreatic cancers with PM. Alternative regimen can be considered multidisciplinary tumour board meeting. Patients will be recruited according to the inclusion criteria and treated for 3 cycles of PIPAC and concurrent systemic chemotherapy. The goal was to repeat PIPAC every 6-8 weeks for at least three procedures, and the delay of the systemic chemotherapy is 2 weeks before and after each PIPAC procedure. If PM was considered to become resectable during PIPAC, patients were discussed at the multidisciplinary tumour board for curative intent cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC). The primary outcome is the clinical benefit rate (CBR), measured by an independent radiologist according to Response Evaluation Criteria In Solid Tumors (RECIST) and Peritoneal Cancer Index (PCI) assessed by laparoscopy and histopathological tumour response evaluated by pathologists blinded to clinical outcomes. Key secondary outcomes include the major and minor treatment-related adverse events according to the Common Terminology Criteria for Adverse Events (CTACE) up to 4 weeks after the treatment, Cytological tumour response of peritoneal lavage or ascites, treatment-related characteristics, hospital stay, progression-free survival, overall survival and readmission rate. The proposed study duration is 3 years from the start date and the estimated sample size is 51 according to centre capacity.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of old;
2. WHO performance of status 0-1;
3. Histologically or cytologically proven PM of a gastric, pancreatic or colorectal carcinoma;
4. Treatment naïve patients as first-line treatment;
5. Progression on or intolerance to first-line systemic chemotherapy as second-line treatment;
6. No symptoms of gastrointestinal obstruction;
7. No contraindications for the planned systemic therapy or laparoscopy;
8. No previous PIPAC/IP/HIPEC;
9. No other concurrent malignancies or any other malignancy within 6 months prior to enrolment;
10. Able to give written informed consent.

Exclusion Criteria:

1. A history of allergic reaction to platinum containing compounds or doxorubicin;
2. Pregnant or breastfeeding;
3. Any extra-peritoneal metastases;
4. Renal impairment, defined as GFR less than 40 mL/min;
5. Impaired liver function defined as bilirubin over 1.5 × UNL;
6. Inadequate haematological function

   * Leucocyte < 3.00 × 109/L
   * Absolute neutrophil counts < 1.50 × 109/L
   * Platelet < 100 × 109/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit rate (CBR) | At the end of Cycle 3 (each cycle is 6 to 8 weeks)
  Clinical benefit rate (CBR) according to Response Evaluation Criteria In Solid Tumors (RECIST).

CONTACTS AND LOCATIONS:
Overall Officials: Ian WONG, Dr., Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No